CLINICAL TRIAL: NCT01203774
Title: "Comparison of SoloSTAR With a Syringe-administered Glargine Insulin in Diabetic Patients Discharged From the Hospital"
Brief Title: Comparison of SoloSTAR With a Syringe-administered Glargine Insulin in Diabetic Patients From the Hospital
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10-0788
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Results first posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pen-administered vs syringe-admnistered Glargine (Active Comparator): SoloSTAR pen-administered Glargine insulin then syringe-administered Glargine insulin
  Interventions: Drug: Glargine insulin
- Syringe-administered vs pen-administered Glargine (Active Comparator): Syringe-administered Glargine insulin and then pen-administered Glargine insulin
  Interventions: Drug: Glargine insulin

INTERVENTIONS:
Drug: Glargine insulin — 20-180 units per day

SUMMARY:
In this study the investigators would like to test the hypothesis that in diabetic patients discharged from the hospital, SoloSTAR Glargine insulin will be superior to syringe-injected Glargine in terms of diabetes control, compliance, and patient satisfaction and preference. The investigators will test this hypothesis in a randomized, crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients with type 1 and 2 diabetes discharged from the hospital with recommendations to take Glargine

Exclusion Criteria:

* Patients unwilling to participate and patients incapable of complying with the study regimen, such as patients with alcohol and drug addiction problems and patients with severe mental illness

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Draznin, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although this is a crossover study, no information is available on the participants that completed phase 1 and started phase 2, and so these milestones are not included. Multiple attempts were made to obtain this information, however the PI is retired and data could not be obtained from any remaining personnel associated with the study. The number of participants started and completed reflects the participants confirmed to have started and completed the study. 43 participants were consented.
Groups:
- Pen-administered, Then Syringe-admnistered Glargine: SoloSTAR pen-administered Glargine insulin then syringe-administered Glargine insulin
  Glargine insulin: 20-180 units per day
- Syringe-administered Then Pen-administered Glargine: Syringe-administered Glargine insulin and then pen-administered Glargine insulin
  Glargine insulin: 20-180 units per day
Period: Overall Study
Arm/Group | Pen-administered, Then Syringe-admnistered Glargine | Syringe-administered Then Pen-administered Glargine
Started | 21 | 10
Completed | 21 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants are grouped into a single arm because no demographics information regarding the separate arms exists. Consented participants that did not complete the study cannot be excluded. Multiple attempts were made to obtain more precise data, however the PI has retired and neither he nor any members of the study team or other contacts associated with the study were able to locate the data.
Groups:
- All Participants: Pen-administered, then syringe-admnistered Glargine Group (1) AND Syringe-administered then pen-administered Glargine Group (2)
  Group 1: SoloSTAR pen-administered Glargine insulin then syringe-administered Glargine insulin Glargine insulin: 20-180 units per day
  Group 2: Syringe-administered Glargine insulin and then pen-administered Glargine insulin Glargine insulin: 20-180 units per day
Arm/Group | All Participants
Number analyzed (Participants) | 43
Age, Customized [Count of Participants; unit: Participants]
  Age 22-70 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: HbA1c at Three Months of Each Period of Treatment
Description: Data was collected by group
Time Frame: Baseline, Month 3 (End of Intervention 1), Month 6 (End of intervention 2)
Population: The only outcome measure available for this measurement is "by group". This measure cannot be entered "by intervention" (e.g. Arm 1: "Pen", Arm 2: "Syringe"). Multiple attempts were made to obtain this information, however the PI is retired and data could not be obtained from any remaining personnel associated with the study. Participants that did not complete the study are not included.
Measure: Mean (Standard Deviation); unit: percentage (DCCT unit)
Groups:
- Group 1: Pen-administered, Then Syringe-admnistered Glargine: SoloSTAR pen-administered Glargine insulin then syringe-administered Glargine insulin
  Glargine insulin: 20-180 units per day
- Group 2: Syringe-administered Then Pen-administered Glargine: Syringe-administered Glargine insulin and then pen-administered Glargine insulin
  Glargine insulin: 20-180 units per day
Arm/Group | Group 1: Pen-administered, Then Syringe-admnistered Glargine | Group 2: Syringe-administered Then Pen-administered Glargine
Number analyzed (Participants) | 21 | 10
percentage (DCCT unit)
  Baseline HbA1c | 10.7 (2.2) | 11.2 (2.5)
  HbA1C at 3 months (end of intervention 1, before crossover) | 7.8 (1.7) | 7.3 (1.4)
  HbA1c at 6 Months (end of dose 2, after crossover) | 8.5 (2.0) | 7.1 (1.6)

2. Secondary Outcome: Compliance and Patient Satisfaction
Time Frame: 6 months of treatment after discharge from the hospital
Population: No data is available for this outcome measure. Multiple attempts were made to obtain this information, however the PI is retired and data could not be obtained from any remaining personnel associated with the study.
Arm/Group | Group 1: Pen-administered, Then Syringe-admnistered Glargine | Group 2: Syringe-administered Then Pen-administered Glargine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Pen-administered Glargine; Syringe-administered Glargine: Glargine insulin: 20-180 units per day
Arm/Group | Pen-administered Glargine | Syringe-administered Glargine
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

LIMITATIONS AND CAVEATS:
Limited results information is available. Multiple attempts were made to obtain this information, however the PI is retired and additional data could not be obtained from any remaining personnel associated with the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No